CLINICAL TRIAL: NCT02260440
Title: A Phase 2 Study of Pembrolizumab (MK-3475) in Combination With Azacitidine in Subjects With Chemo-refractory Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anuradha Krishnamurthy (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Anuradha Krishnamurthy, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-118
Record Dates: First submitted 2014-10-06; First posted 2014-10-09 (Estimated); Results first posted 2017-05-16 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — pembrolizumab; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pembrolizumab and Azacitidine Arm (Experimental): 9 cycles
  * Pembrolizumab will be given at 200 mg every 21 days.
  * Azacitidine will be given at 100 mg daily subcutaneous injection on days 1-5 every 21 days.
  Interventions: Drug: Pembrolizumab; Drug: Azacitidine

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab will be given at 200 mg every 21 days
Drug: Azacitidine — Azacitidine will be given at 100 mg daily subcutaneous injection on days 1-5 every 21 days.

SUMMARY:
This is an open label, single-arm, Phase 2 trial to evaluate the anti-tumor activity, safety, and tolerability of Pembrolizumab in combination with azacitidine in subjects with chemo-refractory mCRC without any further standard treatment options

Dosage and regimen for all study periods

* Pembrolizumab will be given at 200 mg every 21 days.
* Azacitidine will be given at 100 mg daily subcutaneous injection on days 1-5 every 21 days.

The first assessment of tumor response will be performed after cycle 3 (9 weeks), and thereafter approximately every 9 weeks, every 3 cycles of therapy. The modified RECIST 1.1 will be used to establish disease response or progression.

All patients will be evaluated and graded for adverse events according to the NCI Common Terminology for Adverse Events, version 4.0 (NCI-CTCAE).

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Be 18 years of age or older on day of signing informed consent.
3. The diagnosis of mCRC will be based on histologic or cytologic confirmation.
4. Have mCRC that has been previously treated with currently approved standard therapies.
5. Have measurable disease based on RECIST 1.1.
6. At least 1 of the tumor sites must be amenable to core needle biopsy and this may not be the site of disease used to measure antitumor response. Patient must agree to this mandatory biopsy.
7. Have a performance status of 0 or 1 on the ECOG Performance Scale.
8. Demonstrate adequate organ function, all screening labs should be performed within 14 days of treatment initiation.
9. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
10. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
11. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has had a prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
4. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   - Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
5. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy..
6. Has extensive metastatic tumor burden in the liver with serum albumin <3.0 g/dL.
7. Has known renal tubular acidosis with serum bicarbonate <20 mEq/L.
8. Has a known hypersensitivity to azacitidine or mannitol.
9. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment.
10. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study.
11. Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
12. Has an active infection requiring systemic therapy.
13. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
14. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
15. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
16. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
17. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
18. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).

Has received a live vaccine within 30 days prior to the first dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-01; Primary Completion 2016-03 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anuradha Krishnamurthy, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Kuang C, Park Y, Augustin RC, Lin Y, Hartman DJ, Seigh L, Pai RK, Sun W, Bahary N, Ohr J, Rhee JC, Marks SM, Beasley HS, Shuai Y, Herman JG, Zarour HM, Chu E, Lee JJ, Krishnamurthy A. Pembrolizumab plus azacitidine in patients with chemotherapy refractory metastatic colorectal cancer: a single-arm phase 2 trial and correlative biomarker analysis. Clin Epigenetics. 2022 Jan 6;14(1):3. doi: 10.1186/s13148-021-01226-y. PMID 34991708

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab and Azacitidine: 200 mg of Pembrolizumab was administered intravenously over 30 minutes on Day 1 of every 21 day cycle. 100 mg of Azacitidine was given daily via subcutaneous injection on days 1-5 every 21 days.
  Treatment continued for 9 cycles (about 27 weeks) or until there was an evidence of progression of disease (PD) or unacceptable toxicity before the completion of the planned 9 cycles.
Period: Overall Study
Arm/Group | Pembrolizumab and Azacitidine
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab and Azacitidine
Number analyzed (Participants) | 31
Age, Continuous [Median (Full Range); unit: years] | 61 [30 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: The objective response rate is estimated by the proportion (percentage) of participants with the best response of complete response (CR), or partial response (PR) by RECIST 1.1 criteria, with corresponding exact 95% confidence limits being reported. Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 14 months
Population: Participants who received at least one dose of study therapy (median, 3 cycles; range, 1-8).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pembrolizumab and Azacitidine
Number analyzed (Participants) | 30
percentage of participants | 3 [1 to 17]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free Survival (PFS) (median) was determined using the number of months measured from the initial date of treatment to the date of documented progression, or the date of death (in the absence of progression) of participants. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Up to 2 years
Population: Participants who received at least one dose of study therapy (median, 3 cycles; range, 1-8).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab and Azacitidine
Number analyzed (Participants) | 30
months | 2.1 [1.8 to 2.8]

3. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) (median) was determined using the number of months measured from the initial date of treatment to the recorded date of death of participants.
Time Frame: Up to 2 years
Population: Participants who received at least one dose of study therapy (median, 3 cycles; range, 1-8).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab and Azacitidine
Number analyzed (Participants) | 30
months | 6.2 [3.5 to 8.7]

ADVERSE EVENTS:
Arm/Group | Pembrolizumab and Azacitidine
Serious Adverse Events (participants affected / at risk) | 13/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab and Azacitidine (N=30)
Anemia (Blood and lymphatic system disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 2
Death NOS (General disorders) | 1
Fatigue (General disorders) | 1
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1
Rash pustular (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Lethargy (Nervous system disorders) | 1
Stroke (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab and Azacitidine (N=30)
Anemia (Blood and lymphatic system disorders) | 18
Sinus bradycardia (Cardiac disorders) | 3
Diarrhea (Gastrointestinal disorders) | 2
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 9
Fever (General disorders) | 2
General disorders and administration site conditions - Other, specify (General disorders) | 3
Pain (General disorders) | 3
Fatigue (General disorders) | 12
Creatinine increased (Investigations) | 4
Neutrophil count decreased (Investigations) | 4
Platelet count decreased (Investigations) | 4
Blood bilirubin increased (Investigations) | 5
White blood cell decreased (Investigations) | 7
Alanine aminotransferase increased (Investigations) | 9
Lymphocyte count decreased (Investigations) | 9
Aspartate aminotransferase increased (Investigations) | 11
Alkaline phosphatase increased (Investigations) | 14
Anorexia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 4
Hypernatremia (Metabolism and nutrition disorders) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 7
Hyponatremia (Metabolism and nutrition disorders) | 16
Hypoalbuminemia (Metabolism and nutrition disorders) | 18
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes